CLINICAL TRIAL: NCT06371625
Title: Ultrasound Guided Transversus Thoracic and Pectoral Nerve Block Versus Pectoral Nerve Block in Modified Radical Mastectomy
Brief Title: U/S Guided Transversus Thoracic and Pectoral Nerve Block Versus Pectoral Nerve Block in MRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mohamed Soliman (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Soliman, lecturer of anesthesia, National Cancer Institute, Egypt
Organization: National Cancer Institute, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AP2202-30104
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Analgesia
Keywords: Breast Neoplasms; Analgesics; Opioids; Postoperative Pain; Mastectomy; Nerve block
MeSH Terms: conditions — Breast Neoplasms; Agnosia; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: to determine the analgesic effect of ultrasound guided Transversus Thoracic and Pectoral Nerve Block compared to ultrasound guided Pectoral Nerve Block in patients undergoing modified radical mastectomy regarding the following : 1-Post-operative opioid (morphine) consumption in the 1st 24 hours 2- Postoperative Numeric Pain Rating Scale. 3. Effect on hemodynamics: Mean arterial blood pressure and Heart rate. 4. Intraoperative fentanyl consumption. 5. Duration of analgesic effect
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 11 per group. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transeversus Thoracic Plane Block (TTPB) [Group A]: (Active Comparator): block performed in a supine position before general anesthesia. Linear probe of the ultrasound system will be attached at sagittal plane to the sternum and counted from T2 near the clavicle to T5. Then the linear probe will be rotated by 90° and attached between the forth and the fifth costal cartilages connecting at the sternum near nipple. Then, the transversus thoracic muscle and the internal intercostal muscle will be identified.
  Interventions: Procedure: Transeversus Thoracic Plane Block (TTPB) and Pectoral Nerves (PECS) Block
- Pectoral Nerves (PECS) Block [Both Groups] : (Active Comparator): Positioned supine with the ipsilateral arm abducted and externally rotated. The infra-clavicular and axillary regions will be cleaned with chlorhexidine. The probe will be positioned under the lateral third of the clavicle. After locating the subclavian artery, the axillary artery and the axillary vein we will move the probe distally towards the axilla, until the pectorals major muscle is identified. We will start counting the ribs, from 1st rib under the axillary artery and maintaining the pectorals major as a reference, we will move distally and laterally until the lateral border of pectorals major is reached. Serratus anterior muscle cover 2nd, 3rd, 4th rib, this point being the entrance into the anterior axillary line we will use atraumatic needle with extension line and electrode for nerve stimulator (Stimuplex D).
  Interventions: Procedure: Transeversus Thoracic Plane Block (TTPB) and Pectoral Nerves (PECS) Block; Procedure: Pectoral Nerves (PECS) Block

INTERVENTIONS:
Procedure: Transeversus Thoracic Plane Block (TTPB) and Pectoral Nerves (PECS) Block — The TTP block will be performed in a supine position before general anesthesia. First, a high linear probe of the ultrasound system will be attached at sagittal plane to the sternum and counted from T2 near the clavicle to T5. Then the linear probe will be rotated by 90° and attached between the forth and the fifth costal cartilages connecting at the sternum near nipple. Then, the transversus thoracic muscle and the internal intercostal muscle will be identified. A total of 15 mL of 0.25% bupivacaine will be injected into the interfascial plane, between the transversus thoracic muscle and the internal intercostal muscle between the fourth and fifth costal cartilages connecting at the sternum. Pleural downward displacement will be used as an ultrasound endpoint.
Procedure: Pectoral Nerves (PECS) Block — Patients positioned supine with the ipsilateral arm abducted and externally rotated. The infra-clavicular and axillary regions will be cleaned with chlorhexidine. The skin point of and once the structures are identified with ultrasound, the probe will be positioned under the lateral third of the clavicle. After locating the subclavian artery, the axillary artery and the axillary vein we will move the probe distally towards the axilla, until the pectorals major muscle is identified. We will start counting the ribs, from 1st rib under the axillary artery and maintaining the pectorals major. Serratus anterior muscle cover 2nd, 3rd, 4th rib, this point being the entrance into the anterior axillary line we will use atraumatic needle with extension line and electrode for nerve stimulator (Stimuplex D). We will inject 10ml of 0.25% bupivacaine between the pectorals muscles first, then inject 20ml of 0.25% bupivacaine.
  Arms: Pectoral Nerves (PECS) Block [Both Groups] :

SUMMARY:
Interfascial blocks score over regional anesthetic techniques such as Transversus Thoracic Plane Block and Pectoral Nerves (PECS) Block as they have no risk of sympathetic blockade, intrathecal or epidural spread, which may lead to hemodynamic instability and prolonged hospital stay. The transversus thoracic muscle plane block (TTP) block is a newly developed regional anesthesia technique which provides analgesia to the anterior chest wall. First described by Ueshima et al. in 2015, the TTP block is a single-shot nerve block that deposits local anesthetic in the transversus thoracic muscle plane between the internal intercostal and transversus thoracic muscles. TTP block targets the anterior branches of the intercostal nerves (T2-6).

Pectoral plane blocks are recently described . PECS block involves deposition of local anesthetic drug between muscle planes. PECS I block, between Pectoralis Major and Minor at third rib level, and PECS II block, the drug is deposited between Pectoralis minor and Serratus anterior muscle.

The pectoral nerves (PECS) block provides analgesia of the lateral mammary region, the intercostobrachial and lateral cutaneous branches of the intercostal nerves (T2-T6), the medial cutaneous nerve of the arm and forearm, and the long thoracic and thoracodorsal nerves. The modified PECS block produces excellent analgesia and can be used to provide balanced anesthesia.

DETAILED DESCRIPTION:
Background and Rationale:

Breast cancer is one of the common malignancies among women. Surgical resection of the primary tumor with axillary dissection is one of the main modalities of breast cancer treatment. The most common modality for anesthesia is general anesthesia with or without regional blocks. It has been reported that 40% of females report moderate to severe pain in the immediate post-operative period after breast cancer surgery. Acute post-surgical pain leads to delayed discharge from post-operative recovery area, impairs pulmonary and immune functions, increases risk of ileus, thromboembolism, myocardial infarction and may lead to increased length of hospital stay.

It is also an important factor leading to the development of chronic persistent post-operative pain in almost half of the patients. Post-operative pain, stress and use of morphine have been elucidated as factors responsible for increased risk of metastasis. Hence, effective perioperative pain management of patients undergoing breast surgery is essential. Regional blocks have been considered one of the modalities for effective perioperative pain control. They have an opioid-sparing effect and allow early mobilization and early discharge from the hospital.

Interfascial blocks score over regional anesthetic techniques such as Transversus Thoracic Plane Block and Pectoral Nerves (PECS) Block as they have no risk of sympathetic blockade, intrathecal or epidural spread, which may lead to hemodynamic instability and prolonged hospital stay. The transversus thoracic muscle plane block (TTP) block is a newly developed regional anesthesia technique which provides analgesia to the anterior chest wall. First described by Ueshima et al. in 2015, the TTP block is a single-shot nerve block that deposits local anesthetic in the transversus thoracic muscle plane between the internal intercostal and transversus thoracic muscles. TTP block targets the anterior branches of the intercostal nerves (T2-6).

Pectoral plane blocks are recently described . PECS block involves deposition of local anesthetic drug between muscle planes. PECS I block, between Pectoralis Major and Minor at third rib level, and PECS II block, the drug is deposited between Pectoralis minor and Serratus anterior muscle.

The pectoral nerves (PECS) block provides analgesia of the lateral mammary region, the intercostobrachial and lateral cutaneous branches of the intercostal nerves (T2-T6), the medial cutaneous nerve of the arm and forearm, and the long thoracic and thoracodorsal nerves. The modified PECS block produces excellent analgesia and can be used to provide balanced anesthesia.

Study Methodology:

a) Population of the study:

Female patients 20-60 years old undergoing Modified Radical Mastectomy will be enrolled in our study. They will be randomized into two comparable groups:

Group A (patients): They will receive ultrasound-guided Transversus Thoracic Plane Block, Pectoral Nerves (PECS) Block, and General anesthesia.

Group B (patients): Will receive Pectoral Nerves (PECS) Block and General Anesthesia.

Interventions:

* Patient preparation:

All included patients will undergo the following: History taking, physical examination, CBC and coagulation profile. They will be informed about the procedure and its possible complications. Finally, written consent will be taken. They will randomly be allocated into two groups using computer generated random numbers.

Both groups will receive Pectoral Nerves (PECS) Block and General Anesthesia. Group (A) Will have in addition to this anesthesia, Transversus Thoracic Plane Block.

- Procedures: All patients will be kept fasting overnight and will be pre-medicated with midazolam 2mg and 500 ml lactated ringer's solutions will be infused 30 minutes before surgery and will be fully monitored by ECG, blood pressure and pulse oximetry. The ultrasound device (Sonosite M-Turbo C 04TRGD) with a 10-12 MHZ linear array probe (HFL38) will be used.

Group (A): Will receive Transversus Thoracic Plane Block with bupivacaine 0.25% 15ml single injection at same side at T4-T5 level before induction of General Anesthesia. The block will be performed under complete aseptic precautions with a 22 gauge echogenic needle using the same ultrasound machine and linear array probe by an anesthetist not involved in the preoperative assessment of the patient, anesthesia management and data collection.

Group (B): Will receive Pectoral Nerves (PECS) Block and General Anesthesia.

Transeversus Thoracic Plane Block (TTPB) [Group A]:

The TTP block will be performed in a supine position before general anesthesia. First, a high linear probe of the ultrasound system will be attached at sagittal plane to the sternum and counted from T2 near the clavicle to T5. Then the linear probe will be rotated by 90° and attached between the forth and the fifth costal cartilages connecting at the sternum near nipple. Then, the transversus thoracic muscle and the internal intercostal muscle will be identified. A total of 15 mL of 0.25% bupivacaine will be injected into the interfascial plane, between the transversus thoracic muscle and the internal intercostal muscle between the fourth and fifth costal cartilages connecting at the sternum. Pleural downward displacement will be used as an ultrasound endpoint. After the injection, the spread of local anesthetic will be confirmed by using the probe.

Pectoral Nerves (PECS) Block [Both Groups] :

Patients will be positioned supine with the ipsilateral arm abducted and externally rotated. The infra-clavicular and axillary regions will be cleaned with chlorhexidine. The skin point of puncture will be infiltrated with 2% lidocaine and once the structures are identified with ultrasound, the probe will be positioned under the lateral third of the clavicle. After locating the subclavian artery, the axillary artery and the axillary vein we will move the probe distally towards the axilla, until the pectorals major muscle is identified. We will start counting the ribs, from 1st rib under the axillary artery and maintaining the pectorals major as a reference, we will move distally and laterally until the lateral border of pectorals major is reached. Serratus anterior muscle cover 2nd, 3rd, 4th rib, this point being the entrance into the anterior axillary line we will use atraumatic needle with extension line and electrode for nerve stimulator (Stimuplex D). We will use one needle approaches instead of two. We will inject 10ml of 0.25% bupivacaine between the pectorals muscles firstly then inject 20ml of 0.25% bupivacaine between the pectorals major muscle and the serratus muscle. The block will be performed with the patient fully awake, followed by general anesthesia.

Both groups will receive General Anesthesia:

* Induction: propofol 1.5-2mg/kg, fentanyl 1ug/kg and Atracurium 0.5mg/kg.
* Intubation: Endotracheal Intubation with appropriate size.
* Maintenance: Isoflurane, fentanyl and Atracurium (0.1-0.2 mg/kg), according to Train of Four Monitoring. Additional boluses of fentanyl (0.3ug/kg) will be administered to maintain mean arterial blood pressure or heart rate values within 30% of baseline vital signs when the patient entered the operating room. Fentanyl frequency and amount will be documented.
* Monitoring: SPO2, ECG, non-invasive blood pressure (before induction, after tracheal intubation, at skin incision, and then every 5 minutes).
* Maintenance fluids: lactated ringer will be given according to fluid chart maintenance, deficit, third space, and urine output and blood loss.

Methodology:

Age, weight, and duration of Anesthesia will be documented. HR in beats per minute, mean arterial blood pressure (MABP), and ECG changes will be monitored and recorded at the following periods: preoperative, after block, after induction of Anesthesia, at skin incision, and then every 5 min. till the end of the surgery.

Postoperative HR , mean arterial blood pressure ,ECG changes, oxygen saturation of the room air, respiratory rate, assessing pain using VAS score, time to first analgesia request, quantity and frequency of opioid requirements will continuously be monitored and recorded at the following periods: at PACU admission, at 1, 2, 4, 6, 12, and 24 h after surgery at rest., Group (B) will receive Pectoral Nerves (PECS) Block and General Anesthesia).

Sample size:

The aim of this study is to measure the postoperative pain score scale (VAS) in 2 groups of MRM patients (Group A (experimental group) will receive ultrasound guided Transversus Thoracic Plane Block, Pectoral Nerves Block and General anesthesia while Group B (control group) will receive Pectoral Nerves Block and General Anesthesia). Based on a previous study by Ueshima and Otake (2017); the median visual analog scale (VAS) score (in millimetres at rest) at 12 hours postoperatively among the experimental group (who received ultrasound guided Transversus Thoracic Plane Block, Pectoral Nerves Block and General anesthesia) was 14 mm and ranged from (5-18 mm) while the median VAS score at the same time point among the control group (who received Pectoral Nerves Block and General Anesthesia) was 30 mm and ranged from (15-59 mm). A total sample size of 22 MRM patients (11 per group) will be needed for this study with type I error (alpha) 5% and type II error (Beta) 1%. This sample will be increased by 15% (to compensate for non-parametric use) to be 26. To allow for 25% expected losses, the sample will be further increased to 34 MRM patients (17 in each group). Sample size estimation was performed by MedCalc Statistical Software version 14.8.1.

ELIGIBILITY:
Inclusion Criteria:

* female patients.
* type of surgery: MRM
* ASA I, II, III
* BMI >20 kg/m2 and <35 kg/m2

Exclusion Criteria:

* BMI <20 kg/m2 and >35 kg/m2
* known sensitivity or contraindication to drugs used
* history of psychological disorders.
* patient refusal
* pregnancy
* contraindication to regional anesthesia e.g. local sepsis, pre-existing peripheral neuropathy and coagulopathy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | 24 hours postoperatively
  total morphine consumption as iv analgesic

SECONDARY OUTCOMES:
visual analogue scale "VAS score" | 24 hours postoperative
  visual analogue scale as zero "No pain" and 10 "maximum pain"
mean blood pressure | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively
  mean blood pressure changes
heart rate | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively
  heart rate change
first analgesic dose | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively
  time of first analgesic dose

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - National cancer Insititute Cairo university, Cairo
  - National cancer Insititute, Cairo
  - Ahmed Mohamed Soliman, Giza

IPD SHARING:
Plan to Share IPD: Undecided
till publication